CLINICAL TRIAL: NCT03509805
Title: Sleep Apnea Syndrome in Obese Women During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2008_32; 2009-A01018-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-04-24; First posted 2018-04-26 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Apnea, Obstructive Sleep; Pregnancy Complications; Pre-Eclampsia; Obesity
Keywords: sleep apnea syndrome; obesity; pregnancy; preeclampsia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pregnancy Complications; Pre-Eclampsia; Obesity; Sleep Apnea Syndromes | interventions — Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OSA in obese patient during pregnancy (Experimental): OSA in polysomnography
  Interventions: Diagnostic Test: polysomnography
- no OSA in obese patient during pregnancy (Experimental): no OSA in polysomnography
  Interventions: Diagnostic Test: polysomnography

INTERVENTIONS:
Diagnostic Test: polysomnography

SUMMARY:
Excess weight or obesity is associated with an increased risk of health disorders: high blood pressure, diabetes, cardiovascular risks, dyslipidemia and sleep apneas. During pregnancy in obese women, the risk of preeclampsia increases by three and the risk of fetal death in utero by five. Snoring and Obstructive sleep apnea (OSA) may be associated with increased risk of adverse pregnancy outcomes, including maternal cardio pulmonary status, fetal heart rate and fetal acidosis-basis status by recurrent upper-airway obstruction, hypoventilation, and intermittent nocturnal hypoxia. Reports in pregnancy have identified in association with OSA and preeclampsia, intrauterine growth restriction and stillbirth.

The prevalence of OSA among women is estimated to be 2-5%, but it remains underdiagnosed during pregnancy. In sleep apnea syndrome, a few data have shown better pregnancy and fetal outcome with the use continuous positive airway pressure (CPAP) therapy.

the hypothesis is in obese pregnant women that there could be a significant association between sleep apnea syndrome and hypertensive disorders, preeclampsia and adverse fetal outcomes This is a prospective study of Women with a body mass index of 35 kg.m2 or greater. The aim of this study is to determinate the prevalence of sleep apnea syndrome in obese pregnant women and the benefit of CPAP on the maternal and fetal outcome.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* BMI > 35
* > 24th weeks of pregnancy
* informed consent,
* health assurance

Exclusion Criteria:

* no informed consent
* twin pregnancy or more
* no health assurance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnancy
Enrollment: 89 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-03-14 (Actual)

PRIMARY OUTCOMES:
Occurrence of apnea objectified by polysomnography according to specific neurophysiological criteria | during the sleep time, an average 8 hours

SECONDARY OUTCOMES:
occurrence of vascular disease | from inclusion at the beginning of the management of pregnancy to delivery
  High blood pressure (HTAG), Essential or chronic hypertension, preeclampsia, Severe preeclampsia
Evaluation of fetal impact by correlation of birth weight to gestational age | from inclusion at the beginning of the management of pregnancy to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Frédérique Dalmas, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU,Hôpital Jeanne de Flandre, Lille, North, France

IPD SHARING:
Plan to Share IPD: No